CLINICAL TRIAL: NCT02344225
Title: Synergistic Pharmacologic Intervention for Prevention of ROP (SPIPROP STUDY)
Acronym: SPIPROP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: State University of New York - Downstate Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Khadija Sikriti, Clinical Trials Project Manager, State University of New York - Downstate Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 349622; 1U54HD071594 (NIH)
Record Dates: First submitted 2015-01-07; First posted 2015-01-22 (Estimated); Results first posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — caffeine citrate; Caffeine; Ibuprofen; Ketorolac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Caffeine+Saline IV+Saline drops (Active Comparator): Caffeine citrate IV (20 mg/kg loading dose, 5 mg/kg/day maintenance dose) plus placebo saline IV (1 ml/kg followed by 0.25 ml/kg) for 5 days plus sterile normal saline (one drop two times a day) for 14 days (n=40); Caffeine is the intervention
  Interventions: Drug: Caffeine citrate
- Caffeine+Ibp IV+Saline drops (Experimental): Caffeine citrate as described in group 1, plus Ibuprofen (10 mg/kg loading dose followed by low dose ibuprofen 2.5 mg/kg/day) for 5 days plus sterile normal saline (one drop two times a day) for 14 days (n=40); Ibuprofen is the intervention
  Interventions: Drug: Ibuprofen
- Caffeine+Saline+Ketorolac drops (Experimental): Caffeine citrate plus saline IV placebo as described in group 1, and Ketorolac (Acuvail) eye drops (one drop two times a day) for 14 days (n=40); Ketorolac is the intervention
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Caffeine citrate — Caffeine citrate IV (20 mg/kg loading dose, 5 mg/kg/day maintenance dose)
  Other Names: Caffeine
  Arms: Caffeine+Saline IV+Saline drops
Drug: Ibuprofen — Ibuprofen (10 mg/kg loading dose followed by low dose ibuprofen 2.5 mg/kg/day) for 5 days
  Other Names: Neoprofen
  Arms: Caffeine+Ibp IV+Saline drops
Drug: Ketorolac — Ketorolac (Acuvail) eye drops (one drop two times a day) for 14 days
  Other Names: Acuvail
  Arms: Caffeine+Saline+Ketorolac drops

SUMMARY:
Phase 2, open-label, randomized, multi-center studies in infants and premature infants are necessary to determine treatment and preventative strategies for ROP. This study was designed to: a) target infants at the highest risk of ROP in a large number of centers with variable rates of ROP (all stages and severe ROP or stage 3+); and b) assess whether caffeine plus systemic or ophthalmic NSAID will decrease ROP among infants most at risk for ROP. The study is designed to determine whether the novel treatment regimens are safe and potentially effective for ROP prevention and to obtain requisite data for the development of a Phase III efficacy/safety randomized blinded trial. Since caffeine is used extensively in NICUs as standard of care for ELGANs, no placebo group is included.

DETAILED DESCRIPTION:
This study will evaluate the safety, tolerability and PK-PD of, and to compare and contrast, IV Ibuprofen with Caffeine and Ketorolac eye drops with Caffeine in ELGAN infants <28 weeks GA for 14 days duration to treat and preferably prevent ROP associated with prematurity and ELGAN. The specific aims of this trial are:

Aim 1: To establish the synergistic effect of local ophthalmic NSIADs and systemic caffeine as optimal therapies for the attenuation and/or prevention of severe ROP. Hypothesis: Ocular Ketorolac or systemic Ibuprofen potentiated with systemic Caffeine will prevent or diminish the severity of ROP. We will: a) Evaluate the safety, tolerability, and efficacy of early postnatal local ophthalmic NSIADs for prevention of severe ROP in ELGANs. b) Determine the pharmacokinetics, pharmacodymanics and pharmacogenomics of NSAIDs potentiated with caffeine for prevention of ROP.

Aim 2: To identify a "critical" number of arterial oxygen desaturations as a key risk factor for severe ROP.

Hypothesis: A "critical" number of daily arterial oxygen desaturations during the first two weeks of life is a key risk factor for severe ROP. We will: a) Further define the role of VEGF, IGF, MMPs, and ROS in ROP and correlate the levels with the number of arterial oxygen desaturations. b) Establish and identify whether increased serum VEGF in infants with severe ROP is the diffusible isoform VEGF121. This isoform is formed from VEGF proteolysis by plasmin and MMPs. MMPs also cleave Notch/Dll4, which acts as a regulator of VEGF signaling.

Aim 3: To determine whether infants at risk for severe ROP are haploinsufficient for the delta-like ligand 4 (Dll4).

Hypothesis: ELGANs at risk for severe ROP will have different pattern of gene expression specifically related to the Notch signaling pathway, as has been previously shown in animal models. We will: a) Examine cord blood, cord tissue, and placental tissue to compare the gene profile of VEGF and Notch signaling pathways among infants who develop severe ROP and those who do not; and b) Determine whether NSAIDs and/or Caffeine will confer protective benefits on Notch/Dll4 signaling and prevent the development of severe ROP.

This is a phase 2b, randomized, open label, multi-center, safety, tolerability and efficacy study comparing 3 interventions for possible prevention of ROP. The trial will be conducted in at least 8 investigational sites including the Neonatal networks (SUNY Downstate and the Brooklyn-Queens Neonatal Network sites, SUNY Stony Brook), and Miller Children's Hospital, Long Beach, CA. An independent DSMB will assess safety during the study. This study will monitor for safety while on study drug and for 7 days after last dose of drug. An exploratory study to determine the role of pharmacodynamic, drug concentrations (as surrogate of PK profile) and pharmacogenomics will also be conducted in this patient population.

One hundred and twenty preterm infants (<28 weeks gestation; <1250 grams) between 0 and 72 hours of life will be randomized to receive either:

1. Caffeine citrate IV (20 mg/kg loading dose followed by 5 mg/kg/day maintenance dose) plus placebo saline IV (1 ml/kg followed by 0.25 ml/kg) for 5 days plus sterile normal saline (one drop two times a day) for 14 days (n=40);
2. Caffeine citrate as described in group 1 plus Ibuprofen (10 mg/kg loading dose followed by low dose ibuprofen 2.5 mg/kg/day) for 5 days plus sterile normal saline (one drop two times a day) for 14 days (n=40); and
3. Caffeine citrate plus saline IV placebo as described in group 1, and Ketorolac (Acuvail) eye drops (one drop two times a day) for 14 days (n=40)

ELIGIBILITY:
Inclusion Criteria:

* Neonates at high risk for ROP as outlined by the American Academy of Pediatrics, Section on Ophthalmology; American Association for Pediatric Ophthalmology and Strabismus; and American Academy of Ophthalmology (129) will be enrolled. Inclusion criteria are:

  1. all infants with a birth weight of less than 1250 grams;
  2. all infants with a gestational age of 28 weeks or less; and
  3. all infants who required oxygen therapy and ventilator support within the first 2 days of life.

Exclusion Criteria:

* Exclusion criteria are:

  1. major congenital malformations and or chromosomal anomalies including duct-dependent cardiac anomalies;
  2. maternal antenatal NSAID exposure <72 hours before birth;
  3. renal failure or oliguria defined as a urine flow rate <0.5 mL/kg/hour in the 8 hours prior to randomization. Anuria is acceptable if infant is less than 24 hours of life;
  4. platelet count <75,000.mm3;
  5. clinical bleeding such as oozing from puncture sites; and
  6. participation in other clinical drug trials while subject participates in this study and for 7 days after last dose of study drug.

Max Age: 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2015-01-01; Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob V Aranda, MD, PhD, Principal Investigator — SUNY Downstate Medical Center, University Hospital of Brooklyn
Locations (1):
- SUNY Downstate Medical Center/University Hospital of Brooklyn, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started on Jan 01, 2015, and ended on Jun 30, 2018. Ninety-Eight (98) participants have been screened at five study sites. However, only 14 participants were enrolled. The reasons for poor enrollment were mostly due to refusal to participate, and some did not meet the eligibility criteria. All participants completed the study.
Pre-assignment Details: The study screened 98 subjects when most mothers were admitted for preterm labor. They were treated successfully with tocolysis and other clinical managements (e.g. bed rest, magnesium sulfate etc.) which resulted in prolonging the pregnancy beyond 28 weeks at which time they met exclusion criteria and no longer eligible for the study..
Period: Overall Study
Arm/Group | Caffeine+Saline IV+Saline Drops | Caffeine+Ibp IV+Saline Drops | Caffeine+Saline+Ketorolac Drops
Started | 6 | 3 | 5
Completed | 6 | 3 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caffeine+Saline IV+Saline Drops | Caffeine+Ibp IV+Saline Drops | Caffeine+Saline+Ketorolac Drops | Total
Number analyzed (Participants) | 6 | 3 | 5 | 14
Age, Continuous [Mean (Full Range); unit: Gestational Age in Week] | 25.5 [24.7 to 27] | 26.7 [26.7 to 27.8] | 26.6 [24 to 28] | 26.6 [24 to 28]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 7
  Male | 4 | 1 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 2 | 8
  Not Hispanic or Latino | 3 | 0 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 3 | 4
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 2 | 8
Birth Weight (grams) [Mean (Full Range); unit: Grams] — We enrolled all infants with a birth weight of less than 1250 grams
  Grams | 731.7 [665 to 815] | 1119.3 [992 to 1216] | 1020 [685 to 1200] | 917.7 [665 to 1200]

OUTCOME MEASURES:

1. Primary Outcome: Efficacy as Measured by the Number of Participants Presenting With Retinopathy of Prematurity (ROP) and the Rate of Stages/Grade of ROP.
Description: ROP (all grades) will be graded using International ROP Classification and severe ROP (Stage 3+ disease) or need for laser or Avastin The rate of mild (stage 1), moderate (stage 2) and severe ROP (stages >3) will be calculated as the number of infants diagnosed with ROP over the number of infants receiving retinal examinations. The study enrolled only 14 of the projected sample of 120, and the low enrollment did not allow meaningful analyses of efficacy and safety.
Time Frame: 50 weeks PCA +/- 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Caffeine+Saline IV+Saline Drops | Caffeine+Ibp IV+Saline Drops | Caffeine+Saline+Ketorolac Drops
Number analyzed (Participants) | 6 | 3 | 5
Participants
  No ROP | 5 | 3 | 4
  Mild ROP (Stage 1) | 1 | 0 | 0
  Moderate ROP (Stage2) | 0 | 0 | 1
  severe ROP (stages >3) | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: We did not reach the target number of participants needed to measure statistically reliable outcome measure. The secondary outcome measure included Intraventricular hemorrhage (Papile's criteria) and ocular examination for corneal lesions.
Time Frame: Eye examinations was done at standard of care through discharge and once, at 50 weeks PCA. All infants underwent routine eye examination by a pediatric ophthalmologist according to the International Classification for ROP
Measure: Count of Participants; unit: Participants
Arm/Group | Caffeine+Saline IV+Saline Drops | Caffeine+Ibp IV+Saline Drops | Caffeine+Saline+Ketorolac Drops
Number analyzed (Participants) | 6 | 3 | 5
Participants | 0 | 0 | 1

3. Post Hoc Outcome: Length of Hospital Stay
Description: Safety as measured by Length of hospital stay
Time Frame: on average 6 months
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Caffeine+Saline IV+Saline Drops | Caffeine+Ibp IV+Saline Drops | Caffeine+Saline+Ketorolac Drops
Number analyzed (Participants) | 6 | 3 | 5
Days | 126 (30.1) | 74 (9.0) | 68 (21.8)

ADVERSE EVENTS:
Time Frame: The adverse events data were collected over an average of 6 months.
Arm/Group | Caffeine+Saline IV+Saline Drops | Caffeine+Ibp IV+Saline Drops | Caffeine+Saline+Ketorolac Drops
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3 | 2/5
Serious Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 2/5
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caffeine+Saline IV+Saline Drops (N=6) | Caffeine+Ibp IV+Saline Drops (N=3) | Caffeine+Saline+Ketorolac Drops (N=5)
Death (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Apnea (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 2
Bronchopulmonary dysplasia (BPD (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Necrotizing enterocolitis (NEC) (Gastrointestinal disorders) | 0 | 0 | 2
Intraventricular hemorrhage (IVH) (Nervous system disorders) | 0 | 0 | 1
Patent ductus arteriosus (PDA) (Congenital, familial and genetic disorders) | 2 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Caffeine+Saline IV+Saline Drops (N=6) | Caffeine+Ibp IV+Saline Drops (N=3) | Caffeine+Saline+Ketorolac Drops (N=5)
Respiratory Distress Syndrome (RDS) (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 5

LIMITATIONS AND CAVEATS:
We did not reach the target number of participants needed to achieve target power and statistically reliable results. Slow enrollment also causes delayed reporting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-07): https://cdn.clinicaltrials.gov/large-docs/25/NCT02344225/Prot_SAP_000.pdf